CLINICAL TRIAL: NCT05146050
Title: Changes and Influence Factors of Olfactory Function After Chemo-radiotherapy for Locally Advanced Nasopharyngeal Carcinoma: a Prospective Observational Cohort Study
Brief Title: Olfactory Change After Chemo-radiotherapy for Nasopharyngeal Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, Director of the Department of Nasopharyngeal Carcinoma, Sun Yat-sen University
Other Study IDs: 2021-FXY-446
Record Dates: First submitted 2021-11-18; First posted 2021-12-06 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; Olfactory change
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational cohort study aimed to explore the changes of olfactory function at multiple time points from baseline to 1 year after radiotherapy among the local advanced nasopharyngeal carcinoma patients.

DETAILED DESCRIPTION:
Newly-diagnosed patients with stage III or IV non-metastatic Nasopharyngeal Carcinoma (AJCC 8th) will be recruited. Olfactory function of consecutive patients with nasopharyngeal carcinoma was assessed prospectively before treatment and serially up to 1 year after radiotherapy by the Sniffin' Sticks olfactory function test and by The Questionnaire of Olfactory Disorders (QOD) as well as a patient symptom visual analogue scale. The change in olfactory function and it's influence factors in NPC patients who receiving induction chemotherapy with concurrent chemoradiotherapy will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70, regardless of sex.
* Patients with newly histologically confirmed non-keratinizing nasopharyngeal carcinoma, type of WHO II or III, clinical stage III-IVa (according to the 8th American Joint Committee on Cancer [AJCC] edition).
* ECOG (Eastern Cooperative Oncology Group) score: 0-1.
* Patients receiving induction chemotherapy with concurrent chemoradiotherap.
* Patients must sign informed consent and be willing, and well understood the objective and procedure of this study.

Exclusion Criteria:

* Women in pregnancy or lactation.
* Patients who received additional treatment during the observation period due to disease progression.
* Patients with significantly lower heart, liver, lung, kidney and bone marrow function.
* Patient with severe medical condition.
* with a condition that could cause olfactory dysfunction, such as septum deviation, nasal polyposis, nasopharyngeal necrosis, congenital olfactory dysfunction, septum surgery, head trauma, chronic rhinosinusitis, allergic rhinitis, or psychiatric or neurological disorders, such as Parkinson's, MS and Alzheimer's disease, or long history of psychiatric drug, corticosteroids or other drug that may affect olfactory function.
* Not able to return for evaluation of olfactory function or follow-up (language, practical implementation, mental condition)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: nasopharyngeal carcinoma patients
Sampling Method: Non-Probability Sample
Enrollment: 107 (Estimated)
Dates: Start 2021-12-08 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in bjective olfactory function | 1.5 years
  Objective olfactory function was assessed was assessed prospectively before treatment and serially up to 1 year after radiotherapy by TDI-score according to the Sniffin' Sticks olfactory function test.

SECONDARY OUTCOMES:
Change inSubjective olfactory function | 1.5 years
  The Questionnaire of Olfactory Disorders (QOD) will be used during the assessment from baseline to 1 year after radiotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nasopharyngeal Carcinoma, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hua MS, Chen ST, Tang LM, Leung WM. Olfactory function in patients with nasopharyngeal carcinoma following radiotherapy. Brain Inj. 1999 Nov;13(11):905-15. doi: 10.1080/026990599121106. PMID 10579662
- [Background] Ho WK, Kwong DL, Wei WI, Sham JS. Change in olfaction after radiotherapy for nasopharyngeal cancer--a prospective study. Am J Otolaryngol. 2002 Jul-Aug;23(4):209-14. doi: 10.1053/ajot.2002.123436. PMID 12105785
- [Background] Holscher T, Seibt A, Appold S, Dorr W, Herrmann T, Huttenbrink KB, Hummel T. Effects of radiotherapy on olfactory function. Radiother Oncol. 2005 Nov;77(2):157-63. doi: 10.1016/j.radonc.2005.09.015. Epub 2005 Oct 13. PMID 16226328
- [Background] Galletti B, Santoro R, Mannella VK, Caminiti F, Bonanno L, De Salvo S, Cammaroto G, Galletti F. Olfactory event-related potentials: a new approach for the evaluation of olfaction in nasopharyngeal carcinoma patients treated with chemo-radiotherapy. J Laryngol Otol. 2016 May;130(5):453-61. doi: 10.1017/S0022215116000761. Epub 2016 Mar 2. PMID 26931794